CLINICAL TRIAL: NCT06517459
Title: Cultural Modification of an Evidence Based Healthy Lifestyle Intervention for People Post Stroke Who Identify as Hispanic/Latino
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 024-268
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Weight-loss; Stroke; Group Lifestyle Balance; Dietary Behaviors; Physical Activity
MeSH Terms: conditions — Stroke; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the modified GLB-CVA program, available in Spanish or English.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLB CVA Latino (Experimental): The GLB program, adapted for Latino individuals with stroke, will be delivered to participants over a 12-month period, divided into 22 in-person or virtual, group sessions. The goal of the GLB program is to help the participant achieve and maintain a 5-7% weight-loss using a two-pronged approach:
  1. Physical activity: This is based upon recommendations by the American Heart Association and the American College of Sports Medicine (ACSM) to achieve 150 minutes of moderate intensity activity each week. Walking is the primary activity recommended.
  2. Healthy eating: Based on United States Department of Agriculture guidelines, the GLB emphasizes healthy eating patterns and tracking dietary intake. Key recommendations include individuals consuming (1) a variety of vegetables, (2) whole fruits, (3) whole grains, (4) fat-free or low-fat dairy, (5) a variety of lean proteins, and (6) oils at every meal
  Interventions: Behavioral: Group Lifestyle Balance

INTERVENTIONS:
Behavioral: Group Lifestyle Balance — The Group Lifestyle Balance (GLB) program is a self-management intervention that has been shown to result in weight-loss and reduce the risk for Type 2 diabetes through increased physical activity and healthy eating behaviors in the general population. The GLB is a direct adaptation of the Diabetes Prevention Program, both developed at the Diabetes Prevention and Support Center at the University of Pittsburgh. The GLB is designed for delivery in a group-based, community setting,4 and has resulted in weight-loss in a variety of settings, such as community centers, churches, worksites, and healthcare systems.

SUMMARY:
The purpose of this trial is to examine weight loss for Hispanic/Latino people with stroke (CVA) who take part in a healthy lifestyle program that has been culturally modified for Hispanic/Latino people

DETAILED DESCRIPTION:
Weight gain greatly increases the risk of chronic diseases such as diabetes, metabolic syndrome, pulmonary and heart disease. The Group Lifestyle Balance (GLB) intervention is a 12-month, evidence-based weight-loss program that has been used extensively with the general population and with people after CVA, however, it is not adapted to be linguistically and culturally appropriate for Latino persons post stroke. We will modified the program to meet the needs of Latino people with a CVA (GLB-CVA Latino).

Aims:

1. : To create a modification of the CDC-recognized, evidence-based GLB-CVA to be culturally appropriate to meet the unique needs of people who identify as Hispanic/Latino, available in English and Spanish languages, using a Community-Based Participatory Research approach and AB of key stakeholders (patients, caregivers, clinicians, researchers).
2. : Conduct a single-arm trial to describe the effect of participation in the GLB-CVA Latino on primary and secondary outcomes for 24 individuals who identify as Hispanic/Latino (12 English speakers and 12 Spanish speakers) at 3, 6, and 12 months from baseline.
3. : Evaluate the participant compliance (feasibility) and fidelity (adherence to the DPP GLB content) with the GLB-CVA Latino intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25
* Identify as Hispanic or Latino
* 18-85 years of age
* All types of stroke
* Medically able to participate in a weight-loss program
* Physical Activity Readiness Questionnaire +
* ≥12 months post first stroke

Exclusion Criteria:

* Contraindications for physical activity
* Low Cognitive Function
* Residing in hospital, acute rehab, SNF
* Not fluent in English or Spanish
* Pre-existing eating disorder
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | [Time Frame: Baseline, 3, 6, and 12 months]
  Weight will be measured during in-person assessments at BSWIR using a Seca 664 scale. Height will be measured using a stadiometer. Weight and height will be used to calculate BMI. A BodyTrace Smart Scale will be provided to participants to facilitate self-weighing in the home, which include cellular connectivity at no cost to participants so weight will be sent directly to the research team.

SECONDARY OUTCOMES:
HbA1c | [Time Frame: Baseline, 3, 6, and 12 months]
  Fasting venous sample will be obtained for hemoglobin a1c to assess average blood sugar level over the past 2-3 months. Fasting venous samples will also be collected for fasting blood glucose, HDL/LDL, total cholesterol, and triglyceride level. Coordinators are trained phlebotomists
Fasting blood glucose | [Time Frame: Baseline, 3, 6, and 12 months]
  Fasting venous sample will be obtained for hemoglobin a1c to assess average blood sugar level over the past 2-3 months. Fasting venous samples will also be collected for fasting blood glucose, HDL/LDL, total cholesterol, and triglyceride level. Coordinators are trained phlebotomists
Lipid panel | [Time Frame: Baseline, 3, 6, and 12 months]
  Fasting venous sample will be obtained for hemoglobin a1c to assess average blood sugar level over the past 2-3 months. Fasting venous samples will also be collected for fasting blood glucose, HDL/LDL, total cholesterol, and triglyceride level. Coordinators are trained phlebotomists
Circumference | [Time Frame: Baseline, 3, 6, and 12 months]
  Waist circumference measured at the umbilicus and mid-upper arm circumference following ACSM guidelines.
Height | [Time Frame: Baseline, 3, 6, and 12 months]
  Will be collected using a stadiometer and used to calculate BMI
Blood pressure | [Time Frame: Baseline, 3, 6, and 12 months]
  Using an automatic cuff (average of three readings, patient seated) diastolic and systolic scores will be recorded
8-year Diabetes Risk | [Time Frame: Baseline, 3, 6, and 12 months]
  The Framingham Heart Study diabetes risk score83 will be calculated using predictors including age, gender, fasting glucose, BMI, HDL cholesterol and triglyceride levels, blood pressure, and parental history. Risk score calculator and regression model are free and used in GLB weight-loss trials. The age range for this score is 45 years to 64 years, and therefore only individuals within this age will have calculated scores. Furthermore, the minimum cut-off score is 3.
6 Minute Walk Test (6MWT) | [Time Frame: Baseline, 3, 6, and 12 months]
  Assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity.
10 Meter Walk Test (10MWT) | [Time Frame: Baseline, 3, 6, and 12 months]
  Assesses walking speed in (m/s) which is correlated to mobility in the community, capacity to perform ADLs, risk of falls, re-hospitalization, and risk of cognitive decline.
Behavioral Risk Factor Surveillance System (BRFSS) | [Time Frame: Baseline, 3, 6, and 12 months]
  The BRFSS is a state-based system of health surveys that collects information on health risk behaviors, preventative health practices, and health care access primarily related to chronic disease and injury. The GLB-TBI uses the two subscales of Healthy Eating and Physical Activity from the 2017 version of the BRFSS. It consists of 14 items.
Neighborhood Environment Walkability Scale (NEWS) | [Time Frame: Baseline, 3, 6, and 12 months]
  NEWS assesses participants' perception of neighborhood features related to physical activity and grocery shopping, including residential density, land use mix (including both indices of proximity and accessibility), street connectivity, infrastructure for walking/cycling, neighborhood aesthetics, traffic and crime safety, and neighborhood satisfaction.
Short Assessment of Health Literacy | [Time Frame: Baseline, 3, 6, and 12 months]
  Combined word recognition test and comprehension test using multiple-choice questions. Identifies individuals with low health literacy.
Self-Rated Abilities for Health Practice | [Time Frame: Baseline, 3, 6, and 12 months]
  Includes 28 items to assess health behaviors among people with disabilities and yields a total Health Practices Score plus 4 subscale scores (Exercise, Nutrition, Health Practices, and Psychological Well Being). Items are rated on a 5-point scale from 0 'not at all' to 4 'completely.' Scores range from 0-28 with higher scores indicating higher self-efficacy for the health behaviors.
Stroke Impact Scale - Quality of Life | [Time Frame: Baseline, 3, 6, and 12 months]
  Quality of life will be assessed using the Stroke Impact Scale, which assesses 8 dimensions of health-related quality of life specific to people post stroke including subscales (using a 5pt Likert scale) assessing strength, memory and thinking, emotion, communication, activities of daily living, mobility, hand function, and participation/role function.
Change in Exit Survey | [Time Frame: 12 months]
  Participants will be asked to complete an exit survey at the 12-month assessment, asking about experience in, and satisfaction with, the GLB-CVA Latino (including satisfaction and feasibility with modifications and language translation) and suggestions for improvement.
Brief Acculturation Scale for Hispanics | [Time Frame: Baseline, 3, 6, and 12 months]
  4 item language based measure of acculturation for Hispanic populations.
Social Support for Eating Habits | [Time Frame: Baseline, 3, 6, and 12 months]
  Questionnaire that assesses the frequency of support received from others for healthy eating habits over the past 3 months.
Social Support for Physical Activity | [Time Frame: Baseline, 3, 6, and 12 months]
  Questionnaire that assesses the frequency of support received from others for engaging in physical activity over the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Librada Callender, PhD, MPH, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor Institute for Rehabilitation, Dallas, Texas, United States